CLINICAL TRIAL: NCT01204138
Title: Concomitant Use of Apremilast for the Treatment of Active RA Despite TNF-Inhibition and Methotrexate- CATARA
Acronym: CATARA
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: decision of sponsor to withdraw before initiation; 0 patients enrolled
Sponsor: Stanford University (Other)
Collaborators: Celgene Corporation (Industry)
Responsible Party: Principal Investigator, Mark Genovese, Principle Investigator, Stanford University
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: SU-08312010-6811
Record Dates: First submitted 2010-09-10; First posted 2010-09-17 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Arthritis, Rheumatoid
Keywords: RA, treatment, TNF, cytokines
MeSH Terms: conditions — Arthritis, Rheumatoid | interventions — apremilast

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- placebo (Placebo Comparator): Patient randomized to one of two arms, either placebo, or Apremilast
  Interventions: Drug: Placebo
- Apremilast (Active Comparator): Patients randomized to either placebo or apremilast
  Interventions: Drug: Apremilast

INTERVENTIONS:
Drug: Apremilast — Apremilast 30mg BID
  Arms: Apremilast
Drug: Placebo — Placebo BID
  Arms: placebo

SUMMARY:
A Phase II, single institution, double blind, randomized, placebo controlled, cross-over study exploring the safety and efficacy apremilast in patients with active RA with concomitant use of TNF inhibition. Following a screening period, patients with active disease on stable TNF inhibition will be randomized to receive either apremilast or placebo for a period of 12 weeks. At the end of 12 weeks patients will be assessed for efficacy using the ACR responder index looking for a 20% improvement, then all patients initially randomized and treated in a blinded fashion with apremilast will be crossed over to placebo while those patients initially randomized and treated with placebo will be crossed over to apremilast. Patients will be followed for an additional 12 weeks on treatment to assess both safety and efficacy of this combination treatment. Following 24 weeks of active treatment or early termination, patients will undergo a 28 day safety visit.

DETAILED DESCRIPTION:
The primary objective of this study is to evaluate the efficacy of apremilast when used in combination with a background DMARD and TNF inhibition in patients with active RA using the ACR responder index looking for a 20% improvement.

To evaluate the safety and tolerability of apremilast when used in combination with TNF inhibition in patients with active RA.

To evaluate the clinical outcomes in RA using the individual domains of the ACR responder index1 .

To evaluate the clinical outcomes of RA using the Disease Activity Score (DAS28)2 To investigate the effects of apremilast on change in cytokine plasma concentration levels (from baseline to Week 12) and the achievement of an ACR response

ELIGIBILITY:
Inclusion Criteria:

* Understand and voluntarily sign an informed consent form
* 18 years of age at the time of signing the informed consent form.
* Able to adhere to the study visit schedule and other protocol requirements
* Must have a diagnosis of RA of at least 6 months duration based on the ACR criteria
* Must have evidence of active disease with DAS-28 > 3.8
* May be on one of the following DMARDs for at least 12 weeks and at a stable dose for at least 6 weeks:

  * Methotrexate 7.5-25mg/week
  * Hydroxychloroquine (200-400mg/day)
* Must be on one of the following SQ TNF inhibitors at a stable, label approved dose for at least 12 weeks:

  * adalimumab (Humira®, Abbott Laboratories, North Chicago, IL)
  * certolizumab pegol (Cimzia®, UCB, Inc, Smyrna, GA)
  * golimumab (Simponi®, Johnson & Johnson, New Brunswick, NJ)
  * etanercept (Enbrel®, Amgen, Thousand Oaks, CA and Wyeth Pharmaceuticals, Philadelphia, PA)
* Concommitant use of non-steroidal anti-inflammatory drugs and/or oral corticosteroids (prednisone<10mg/day or equivalent) are permitted if doses have been stable for at least 14 days.
* If taking methotrexate, patient must also be taking folic or folinic acid at at dose of no less then 5mg/week.
* Must meet the following laboratory criteria:

  * Hemoglobin > 9 g/dL
  * White blood cell (WBC) count; 3000 /;L (3.0 X 109/L) and 14,000/L (< 14 X 109/L)
  * Platelets; 100,000 /L (100 X 109/L)
  * Serum creatinine; 1.5 mg/dL (or 133mol/L)
  * Total bilirubin; 2.0 mg/dL
  * Aspartate transaminase (AST [serum glutamic oxaloacetic transaminase, SGOT]) and alanine transaminase (ALT [serum glutamate pyruvic transaminase, SGPT]); 1.5x upper limit of normal (ULN)
* Females of childbearing potential (FCBP)‡ must have a negative urine pregnancy test at screening (Visit 1). In addition, sexually active FCBP must agree to use TWO of the following adequate forms of contraception while on study medication: oral, injectable, or implantable hormonal contraceptives; tubal ligation; intrauterine device; barrier contraceptive with spermicide; or vasectomized partner while on study. A FCBP must agree to have pregnancy tests every 4 weeks while on study medication and for one month after taking the last dose of study medication.
* Males (including those who have had a vasectomy) must agree to use barrier contraception (latex condoms) when engaging in reproductive sexual activity with FCBP while on study medication and for 28 days after taking the last dose of study medication

Exclusion Criteria:

* Inability to provide voluntary consent
* Any condition, including the presence of laboratory abnormalities, which places the subject at unacceptable risk if he/she were to participate in the study or confounds the ability to interpret data from the study
* Pregnant or breastfeeding
* Systemic fungal infection
* Active tuberculosis or a history of incompletely treated tuberculosis
* History of recurrent bacterial infection (at least 3 major infections resulting in hospitalization and/or requiring intravenous antibiotic treatment within the past 2 years)
* Clinically significant abnormality on the chest x-ray (CXR) with anteriorposterior and lateral views at screening. Chest x-rays performed within 3 months prior to start of study drug are acceptable.
* Use of any investigational medication within 4 weeks prior to start of study drug or 5 pharmacokinetic/pharmacodynamic half-lives (whichever is longer)
* Any clinically significant abnormality on 12-lead ECG at screening
* History of congenital or acquired immunodeficiency (eg, Common Variable Immunodeficiency [CVID])
* Hepatitis B surface antigen positive or Hepatitis B core antibody positive at screening
* History of Human Immunodeficiency Virus (HIV) infection
* Antibodies to Hepatitis C at screening
* History of malignancy within 5 years prior to the screening visit (except for treated [i.e. cured] basal cell skin carcinomas and treated [i.e. cured] carcinoma in situ of the cervix)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2010-09; Primary Completion 2011-08 (Actual); Study Completion 2011-12 (Actual)

PRIMARY OUTCOMES:
20% improvement based on ACR responder criteria | 12 weeks

SECONDARY OUTCOMES:
ACR 50/70 and DAS | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Mark Genovese, Principal Investigator — Stanford University
Locations (1):
- Stanford University School of Medicine, Stanford, California, United States